CLINICAL TRIAL: NCT05954975
Title: Objective Assessment of Illness Severity of Infants Presented at the Emergency General Practitioner Post
Brief Title: Baby Sickness Evaluation
Acronym: BeSurE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ilona C Narayen, MD pHD (Other)
Responsible Party: Sponsor-Investigator, Ilona C Narayen, MD pHD, Pediatrician and principal investigator Ilona Narayen, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Other Study IDs: 132698
Record Dates: First submitted 2023-06-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Infant, Newborn, Diseases
Keywords: Screening; BabyCheck; Pulse oximetry; Young infant
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants up to 6 months of age: Infants up to six months of age, presenting with systemic illness at the emergency GP post.
  Interventions: Combination Product: BabyCheck and pulse oximetry

INTERVENTIONS:
Combination Product: BabyCheck and pulse oximetry — The BabyCheck is a validated scoring system to grade the severity of acute systemic illness in infants up to six months of age. Severity of illness is graded by using a weighted score of a combination of nineteen signs and symptoms. The higher the score, the higher the chance of severe illness.
  Nellcor PM10N is a pulse oximeter which is cleared for use in young infants. A sensor for infants will be used, so reliable oxygen saturation and heart rate can be obtained.

SUMMARY:
The goal of this prospective single center feasibility study is to assess the feasibility of using BabyCheck and PO by GPs as an illness severity score for young infants > 6 months of age in order to aid the decision for referral to hospital.

The emergency GP posts in Leiderdorp will add the BabyCheck and PO to their standard evaluation of infants presenting with systemic illness < six months of age for a period of six months.

The feasibility will be determined by calculating the percentage of eligible infants in whom a complete BabyCheck score and PO data were retrieved. The investigators consider the protocol feasible if this is done in 80% of all eligible infants.

DETAILED DESCRIPTION:
Young infants frequently visit general practitioners (GP) with acute pathology, such as infections. Assessing severity of illness in this group is often challenging, since the likelihood of serious illness in this group is low, deterioration of the clinical condition can occur more rapidly. Therefore, early recognition of pathology in young babies is pivotal.

The Netherlands Triage System (derived from the Manchester Triage System) is a reliable tool for both children and adults to decide if a patient should be seen by the GP. However, after presentation at the GP, a scoring system to assess illness severity in babies with a decision aid for referral to hospital, is currently lacking.

The BabyCheck is a scoring system developed and validated as a clinical checklist to assess young infants up to six months of age. The BabyCheck is validated in multiple low illness prevalent settings.

In addition, abnormal oxygen saturation and/or heart rate can be an early sign of infection, respiratory or circulatory pathology in infants. Since it is difficult to adequately judge oxygen saturation solely by skin colour, it is preferable to objectify this parameter via pulse oximetry (PO).

The aim of this study is to assess the feasibility of using BabyCheck and PO by GPs as an illness severity score for young infants < six months of age in order to aid the decision for referral to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Infants up to six months of age.
* Presenting with systemic illness (no injuries or traumata).
* Presenting at the emergency GP post of Leiderdorp.

Exclusion Criteria:

* Infants up to six months of age, presenting with traumata or that are in a resuscitation setting.
* Infants with referral to other hospitals than the Alrijne hospital. The location for referral is coded and available from the anonymized database of the emergency GP post.
* Infant < 1 month of age presenting with fever (body temperature > 38.0 ⁰C), with or without unknown origin, since these infants should always be referred according to the national guidelines for GPs.
* Infants < 3 months of age presenting with fever of unknown origin (temperature > 38.0 ⁰C), since these infants should always be referred according to the national guidelines for GPs.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: Our study population consists of infants up to six months of age, presenting with systemic (non-traumatic/surgical) illness at the emergency GP post.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 6 months
  Feasibility will be determined by calculating the percentage of eligible infants in whom a complete BabyCheck score and PO data were retrieved. We consider the protocol feasible if this is done in 80% of all eligible infants.

SECONDARY OUTCOMES:
Sensitivity and specificity of the combined BabyCheck-PO score | 6 months
  a referral to the pediatric department is assigned just if no treatment, diagnostic tools or follow up is performed in hospital, which could not have been performed at the GP post.
Acceptability of GPs | 6 months
  1. Was the combination of questions and pulse oximetry useful for assessing illness severity in this infant? [yes/no]
  2. Did the outcome of the scores influence your decision for referral? [yes/no]
  3. Do you have any comments for the reseaerchers? [open field]
Acceptability of pediatricians | 6 months
  1. Was the referral necessary or just? [yes/no]
  2. Was the referral possibly previously missed or too much delayed? [yes/no].
  3. Was the combination of BabyCheck and pulse oximetry useful in assessing illness severity in this infant? [yes/no]

IPD SHARING:
Plan to Share IPD: Undecided